CLINICAL TRIAL: NCT02187354
Title: An Open-Label, Multi-center, Expanded Access Protocol of Blinatumomab for the Treatment of Pediatric and Adolescent Subjects With Relapsed and/or Refractory B-precursor Acute Lymphoblastic Leukemia (ALL)
Brief Title: Expanded Access Protocol - Blinatumomab in Pediatric & Adolescent Subjects With Relapsed/Refractory B-precursor ALL
Acronym: RIALTO
Status: No longer available | Type: Expanded Access
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Other Study IDs: 20130320; 2014-001700-21 (EudraCT Number)
Record Dates: First submitted 2014-07-09; First posted 2014-07-11 (Estimated); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Relapsed/Refractory B-Precursor Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Recurrence | interventions — blinatumomab

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Drug: Blinatumomab — A single cycle of blinatumomab (CIVI) treatment is 6wks, 4wks of treatment followed by a 2wk treatment-free interval. Up to 5 cycles will be administered per subject. In the first cycle, for patients with an M3 bone marrow, the initial dose will be 5μg/m2/day for the first 7days, escalated to 15μg/m2/day on D8-D29. For all subsequent cycles 15μg/m2/day will be the dose for all 4wks of continuous treatment. In case of M2 bone marrow or M1 bone marrow with an MRD relapse at screening, the initial dose will start at 15μg/m2/day for the first 7days of treatment & no dose step at D8. For all subsequent cycles the dose will remain 15μg/m2/day. A dose of 9μg/day for the initial dose (if applicable) & 28μg/day for the escalated dose after dose step should not be exceeded.
  Other Names: AMG103, Blincyto
Other: Extension of LTFU as per ProtocolAmendment7 7Jun18 — LTFU (Long Term Follow-Up) will extend past 18 months for patients already ended the study/still on study or to be enrolled at European sites if they did not receive a transplantation after blinatumomab treatment. For subjects to be included in the additional LTFU, data will be captured until subjects are 18yrs old (every 6 months by phone contact). The following will be captured: relapse (medullary or extra-medullary relapse and its specific location), second tumor (which type), alive/died and cause of death, hospitalization and reason for hospitalization.

SUMMARY:
Primary Objective:

To estimate the incidence of treatment-emergent and treatment-related adverse events during treatment with blinatumomab in pediatric and adolescent subjects with B-precursor ALL in second or later bone marrow relapse, in any marrow relapse after alloHSCT, or refractory to other treatments

Secondary Objective(s):

To describe key efficacy outcomes, including incidence of complete response (CR) within 2 cycles of blinatumomab, minimal residual disease (MRD) remission within 2 cycles of blinatumomab, relapse free survival (RFS), overall survival (OS), incidence of alloHSCT, and 100-day mortality after alloHSCT.

Hypotheses:

A formal statistical hypothesis will not be tested. The incidence of treatment-emergent and treatment-related adverse events will be estimated.

Study Endpoints:

* Incidence of treatment-emergent and treatment-related adverse events
* Incidence of CR within 2 cycles of blinatumomab
* MRD remission within 2 cycles of blinatumomab
* RFS
* OS
* Incidence of alloHSCT
* 100-day mortality after alloHSCT

Study Design:

Multi-center, open-label, single-arm expanded access protocol

ELIGIBILITY:
Inclusion Criteria 101 Immunophenotypic evidence of CD19 positive B-precursor ALL (pro B-, pre B-, common ALL) 102 Age > 28 days and < 18 years at the time of informed consent/assent 103 Morphological or molecular evidence of relapsed/refractory disease, defined as one of the following:

* Second or later bone marrow relapse (defined as M3 marrow or M2 marrow or M1 marrow but with MRD level ≥ 10E-3), or
* Any marrow relapse after alloHSCT (defined as M3 marrow or M2 marrow or M1 marrow but with and MRD level ≥ 10E-3), or
* Refractory to other treatments:

  * For patients in first relapse: failure to achieve a CR following a full standard reinduction chemotherapy regimen
  * For patients who have not achieved a first remission: failure to achieve remission following a full standard induction regimen
* Subjects previously treated with blinatumomab may be eligible, if subject ended treatment for reason(s) other than disease progression or intolerability to blinatumomab (Note: This does not include patients who have already received blinatumomab treatment on this study, but refers only to patients outside of the 20130320 study)

Other Inclusion Criteria may apply

Exclusion Criteria 201 Any active acute Graft-versus-Host Disease (GvHD) grade 2 to grade 4 according to the Glucksberg criteria or active chronic GvHD requiring systemic treatment 202 Immunosuppresive agents to prevent or treat GvHD within 2 weeks prior to blinatumomab treatment (except for topical corticosteroids) 203 Active (overt) ALL in the CNS (confirmed by cerebrospinal fluid [CSF] analysis) or in testes

Other Exclusion Criteria may apply

Ages: 0 Years to 17 Years | Sex: All
Age Groups: Child

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (19):
- United States (4):
  - Research Site, Aurora, Colorado
  - Research Site, Cincinnati, Ohio
  - Research Site, Memphis, Tennessee
  - Research Site, Salt Lake City, Utah
- Research Site, Vienna, Austria
- France (2):
  - Research Site, Marseille
  - Research Site, Paris
- Germany (7):
  - Research Site, Berlin
  - Research Site, Frankfurt am Main
  - Research Site, Kiel
  - Research Site, München
  - Research Site, Münster
  - Research Site, Tübingen
  - Research Site, Würzburg
- Italy (3):
  - Research Site, Monza (MB)
  - Research Site, Padua
  - Research Site, Roma
- Research Site, Zurich, Switzerland
- Research Site, Sheffield, United Kingdom

REFERENCES:
- [Background] Locatelli F, Zugmaier G, Mergen N, Bader P, Jeha S, Schlegel PG, Bourquin JP, Handgretinger R, Brethon B, Rossig C, Kormany WN, Viswagnachar P, Chen-Santel C. Blinatumomab in pediatric relapsed/refractory B-cell acute lymphoblastic leukemia: RIALTO expanded access study final analysis. Blood Adv. 2022 Feb 8;6(3):1004-1014. doi: 10.1182/bloodadvances.2021005579. PMID 34979020
- [Background] Locatelli F, Zugmaier G, Mergen N, Bader P, Jeha S, Schlegel PG, Bourquin JP, Handgretinger R, Brethon B, Rossig C, Chen-Santel C. Blinatumomab in pediatric patients with relapsed/refractory acute lymphoblastic leukemia: results of the RIALTO trial, an expanded access study. Blood Cancer J. 2020 Jul 24;10(7):77. doi: 10.1038/s41408-020-00342-x. No abstract available. PMID 32709851
- [Background] Queudeville M, Stein AS, Locatelli F, Ebinger M, Handgretinger R, Gokbuget N, Gore L, Zeng Y, Gokani P, Zugmaier G, Kantarjian HM. Low leukemia burden improves blinatumomab efficacy in patients with relapsed/refractory B-cell acute lymphoblastic leukemia. Cancer. 2023 May 1;129(9):1384-1393. doi: 10.1002/cncr.34667. Epub 2023 Feb 24. PMID 36829303
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com